CLINICAL TRIAL: NCT01543464
Title: Combination of IDO/Survivin Peptide Vaccine, GM-CSF, Imiquimod and Temozolomide Chemotherapy for Patients With Metastatic Malignant Melanoma
Brief Title: Peptide Vaccine and Temozolomide for Metastatic Melanoma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Diminished rectruitment
Sponsor: Inge Marie Svane (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, MD, PhD & Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM1120
Record Dates: First submitted 2012-02-08; First posted 2012-03-05 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Malignant Melanoma
Keywords: Indeolamine 2,3 dioxygenase; Survivin; Montanide; Imiquimod; GMCSF
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine+adjuvants+temozolomide treatment (Experimental): Experimental arm
  Interventions: Drug: Chemotherapy: Temozolomide

INTERVENTIONS:
Drug: Chemotherapy: Temozolomide — Vaccine: 250 microgram IDO5 peptide + 250 microgram Survivin peptide + 500 microL Montanide every 2nd week Adjuvants: 75 microgram GM-CSF + 1 application Imiquimod every 2nd week

SUMMARY:
The aim of the study is to assess if treatment with IDO/Survivin peptide vaccine can enhance the efficacy of temozolomide chemotherapy in patients with metastatic malignant melanoma.

DETAILED DESCRIPTION:
Secondarily to studying the efficacy of the treatment; the investigators examine if treatment with IDO/Survivin peptide can induce a measurable cellular T-cell response when the vaccine is given in combination with temozolomide treatment for melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histological verified malignant melanoma
2. Metastatic disease (brain metastasis allowed if asymptomatic)
3. Evaluable disease recording to RECIST v. 1.1
4. Age > 18 years
5. Performance status, PS=0, PS=1 or PS=2
6. Life expectancy > 3 months
7. Adequate bone marrow function
8. Leucocyte count > 2,5 * 109/L
9. Granulocyte count > 1,5 * 109/L
10. Thrombocyte count > 100 * 109/l
11. Creatinine < 2,5 * UNL 130 micromol/L
12. Adequate liver function
13. ASAT < 100 U/L
14. Bilirubin < 300 U/L
15. S-hCG negative (fertile women)
16. Written informed consent
17. Inclusion at least 4 weeks after major abdominal surgery
18. If radiotherapy for brain metastases prior to inclusion, then progressive disease proven by new brain MR-scan before inclusion

Exclusion Criteria:

1. Treatment with immune suppressors (ie. prednisone) not allowed
2. Other malignancies 3 years prior to inclusion except benign skin lesions
3. Severe medical condition, severe asthma, severe COL, severe heart- or diabetic disease
4. Acute/Chronic infection with HIV, hepatitis or tuberculosis
5. Known severe allergic reactions
6. Former anaphylactic reactions
7. Active autoimmune diseases
8. Pregnant or nourishing women
9. Psychiatric disease resulting in non-compliance
10. Known allergic reactions towards Montanide, Imiquimod, Temozolomide or Leukine
11. Simultaneously treatment with other experimental drugs

Patients cannot be treated with chemotherapy, radiotherapy (except locally) or immunotherapy 14 days within inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR) | 18 months
  Primary endpoint is clinical benefit rate defined as complete remission rate + partial response + stable disease for a minimum of 6 months plus assessment of time to progression (TTP).

CONTACTS AND LOCATIONS:
Overall Officials: Trine Zeeberg Iversen, MD, Principal Investigator — Center for Cancer ImmuneTherapy; Inge Marie Svane, MD, PhD, Prof., Study Director — Center for Cancer ImmunoTherapy
Locations (1):
- Trine Zeeberg Iversen, Brønshøj, Copenhagen, Denmark